CLINICAL TRIAL: NCT04475783
Title: Head-to-Head Comparison of SIROlimus Versus Paclitaxel Drug-Eluting BallooN Angioplasty in the Femoropopliteal Artery
Brief Title: Sirolimus- vs. Paclitaxel-Drug Coated Ballons in Patients With Peripheral Artery Disease
Acronym: SIRONA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Collaborators: Concept Medical Inc. (Industry); Vascuscience (Unknown); CoreLab Black Forest (Unknown); Center for Clinical Studies, Jena University Hospital (Unknown)
Responsible Party: Principal Investigator, Ulf Teichgräber, Prof. Dr., Jena University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZKSJ0127; DRKS00022452 (Other: German Registry for Clinical Trials)
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Artery Disease; Sirolimus; Paclitaxel; Drug-Coated Balloon; Percuteanous Transaluminal Angioplasty; PPA; SFA; MagicTouch PTA
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty

STUDY DESIGN:
Intervention Model Description: 1:1-randomization, parallel design, stratified by Center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sirolomus DCB group (Experimental): Intervention with Sirolimus-coated balloon catheter
  Interventions: Combination Product: Percutaneous Transluminal Angioplasty (PTA)
- Paclitaxel DCB group (Active Comparator): Intervention with Paclitaxel-coated balloon catheter
  Interventions: Combination Product: Percutaneous Transluminal Angioplasty (PTA)

INTERVENTIONS:
Combination Product: Percutaneous Transluminal Angioplasty (PTA) — PTA with an drug-coated balloon catheter (DCB) in the femoropopliteal artery

SUMMARY:
This study is a prospective, interventional, multi-center 1:1 randomized non-inferiority trial.

The trial evaluates the safety and efficacy of the Magic Touch PTA sirolimus drug-coated balloon in comparison to the treatment with PTX drug-coated balloon (control device) in patients with femoropopliteal artery disease.

DETAILED DESCRIPTION:
Percutaneous transluminal angioplasty (PTA), in which a balloon is advanced and inflated in the obstructed artery for several seconds to minutes, has become the standard endovascular treatment for peripheral arteries. The long-term success of bare balloon PTA in the fem-oropopliteal segment is hampered by the occurrence of restenosis, which can be reduced by local antiproliferative drug delivery via the PTA balloon catheter.

The rationale of this study is based on the hypothesis that the usage of the Sirolimus-coated Magic Touch Sirolimus DCB is at least equal (non-inferior) with regards to efficacy and safety in comparison with a clinically well-established PTX coated balloon.

The objective of this prospective, randomized, multi-center, post-market study is to compare the Magic Touch Sirolimus DCB with Paclitaxel-coated DCB for treatment of high grade ste-notic or occluded lesions in SFA and / or P1 segment of the popliteal artery (PA) in PAD pa-tients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age ≥ 18
2. Subject has been informed on the nature of the study, the duration of the study, agrees to attend follow-up visits, agrees to complete the required testing, agrees to participate, and has signed an informed consent form.
3. Rutherford category 2-4 according to the investigator's subjective evaluation
4. Subject has a de novo or re-stenosed lesion with ≥ 70 % stenosis documented angiographically
5. Target lesion length is ≥ 2 cm and ≤ 20 cm by visual estimate of the treating physician
6. Multiple lesions with max. 3 cm healthy vessel segment in between lesions can be considered at the discretion of the operator as one lesion. Total lesion length should not exceed 20 cm
7. Reference vessel diameter (RVD) ≥ 4 mm and ≤ 6.5 mm by visual estimation
8. Patency of P2 and P3 segment of the popliteal artery and at least one (1) infrapopliteal artery to the ankle (< 50 % diameter stenosis) in continuity with the femoropopliteal artery
9. Patency of ipsilateral iliac artery (≤ 30% diameter stenosis). Iliac artery stenosis > 30 % may be treated during the index procedure to ensure sufficient inflow.
10. A guidewire has successfully traversed the target treatment segment intraluminal
11. Vascular disease in the opposite leg that requires treatment at the time point of index procedure is allowed, but has to be treated according to randomization or with POBA.
12. A patient can only be enrolled and randomized once with only one target lesion in the SIRONA trial. Please note that only the lesion in one limb can be treated as target lesion for index procedure.

Exclusion Criteria:

1. Failure to successfully cross the target lesion or subintimal target lesion guidewire crossing
2. Flow-limiting dissection after pre-dilatation
3. Angiographic evidence of severe calcification of the target vessel (contiguous calcification on both sides of the vessel)
4. Presence of fresh thrombus in the target lesion
5. Presence of aneurysm in the target vessel/s
6. Prior vascular surgery (including atherectomy, bypass surgery) of the target limb
7. Prior stent in the target lesion
8. Stroke or heart attack within 3 months prior to enrollment
9. Any vascular surgical procedure or intervention performed in the target limb within 30 days prior to or planned within 30 days post index procedure
10. Any vascular treatment with PTX or sirolimus-coated devices 60 days prior to index procedure
11. Target lesion requires treatment with alternative therapies such as primary stenting, laser, lithotripsy, thrombectomy, atherectomy, cryoplasty, brachytherapy, re-entry devices
12. Enrolled in another investigational drug, device or biologic study
13. Life expectancy of less than one year in the investigator's opinion
14. Known allergies or sensitivity to heparin, aspirin, other anticoagulant/ antiplatelet therapies, sirolimus, paclitaxel or contrast media that cannot be adequately pre-treated prior to index procedure
15. Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy
16. Receiving dialysis or immunosuppressant therapy
17. Pregnant or lactating females
18. History of major amputation in the same limb as the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Patency rate (Absence of clinically driven target lesion revascularization) | one year after study procedure (PTA with medical product under investigation or comparator)
  patency rate after one year defined as absence of clinically driven target lesion revascularization (TLR) due to symptoms and drop of ABI of ≥ 20% or > 0.15 when compared to post-procedure or restenosis with PVR > 2.4 evaluated by duplex ultrasound
Safety outcome | through 12 months post-procedure
  Composite of freedom from device and procedure-related death through 12 months post procedure as well as freedom from both target limb major amputation and clinically-driven target vessel vessel revasculariza-tion

SECONDARY OUTCOMES:
TLR rate | 1, 6, 12, 24, 36, 48 and 60 months after study procedure
  ocurrence of Target lesion revascularization (TLR) at certain time Points
Rutherford classification | at 12 months after study procedure
  Sustained clinical improvement: an improvement shift in the Rutherford classification of one class in amputation and TVR free surviving patients
Walking capacity assessment 1 | at 1, 6, 12, 24, 36, 48 and 60 months after study procedure
  patient-self-assessment of walking distance
Walking capacity assessment 2 | at 6, 12, 24, 48 months after study procedure
  6-minute Walking test (6MWT)
Walking capacity assessment 3 | at 6, 12, 24, 48 months after study procedure
  Treadmill test (optional)
Walking capacity assessment 4 | at 6, 12, 24, 48 months after study procedure
  Walking Impairment Questionnaire (WIQ); 20 questions (scale 0 to 4); best score 0, worst score 80
Duplex Ultrasound | post-procedure and at 6, 12, 24 and 48 months or at any time of re-intervention
  Duplex-defined binary restenosis (PSVR >2.4) of the target lesion
ABI | at discharge, 6, 12, 24 and 48 months
  Ankle brachial index (ABI)
Qualilty of Life Assessment | at 1 month, 6, 12, 24, 36, 48 and 60 months
  Quality of life assessment (QoL) by EQ5D-3L questionnaire; 5 questions (scale 1 to 5), best score 5, worst score 25
Secondary Safety: freedom from all cause death, target limb major amputation and clinically-driven target vessel revascularization | trough 60 months after study procedure
  Composite of freedom from all cause death through 60 months post procedure as well as freedom from both target limb major amputation and clinically-driven target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Teichgraeber, Prof. Dr., Study Director — University Hospital Jena, Institute of Radiology
Locations (22):
- Austria (5):
  - Medical University Vienna, Universitätsklinik für Innere Medizin II, Klinische Abteilung für Angiologie, Vienna, Vienna
  - Medizinische Universität Graz, Klinische Abteilung für Angiologie, Graz
  - Klinikum Klagenfurt am Wörthersee, Institut für Diagnostische und Interventionelle Radiologie, Klagenfurt
  - Universitätsklinik für Radiologie und Nuklearmedizin, Klinische Abteilung für Kardiovaskuläre und Interventionelle Radiologie, Vienna
  - Hanusch-Krankenhaus, Vienna
- Germany (17):
  - University Heart Center Freiburg-Bad Krozingen, Bad Krozingen
  - Fürst-Stirum-Klinik Bruchsal, Klinik für Kardiologie, Angiologie, Diabetologie, Neurologie und Intensivmedizin, Bruchsal
  - Sana Kliniken Oberfranken Coburg, Coburg
  - Universitätsklinikum Dresden, Institut und Poliklinik für Diagnostische und Interventionelle Radiologie, Dresden
  - Universitätsklinikum Essen, Westdeutsches Herz- und Gefäßzentrum Essen, Klinik für Kardiologie und Angiologie, Essen
  - DIAKO Krankenhaus gGmbH, Institut für Diagnostische und Interventionelle Radiologie und Neuroradiologie, Flensburg
  - Universitätsklinikum Heidelberg, Medizinische Klinik III, Kardiologie, Angiologie und Pneumologie, Heidelberg
  - Klinikverbund Allgäu gGmbH, Herz- und Gefäßzentrum Oberallgäu Kempten, Klinik Immenstadt, Immenstadt im Allgäu
  - University Hospital Jena, Jena
  - Helios Klinikum Krefeld, Institut für Diagnostische und Interventionelle Radiologie, Krefeld
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Angiologie, Leipzig
  - Marienhaus Klinikum Mainz, Klinik für Diagnostische und Interventionelle Radiologie, Mainz
  - St. Franziskus-Hospital GmbH, Klinik für Gefäßchirurgie, Münster
  - Universitätsklinikum Münster, Klinik für Kardiologie I, Koronare Herzkrankheit, Herzinsuffizienz und Angiologie, Münster
  - Elblandklinikum Radebeul, Gefäßzentrum, Radebeul
  - Schön Klinik Rendsburg, Institut für Diagnostische und Interventionelle Radiologie/Neuroradiologie, Rendsburg
  - Kreiskrankenhaus Torgau, Abt. Innere Medizin / Angiologie, Torgau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teichgraber U, Ingwersen M, Platzer S, Lehmann T, Zeller T, Aschenbach R, Scheinert D. Head-to-head comparison of sirolimus- versus paclitaxel-coated balloon angioplasty in the femoropopliteal artery: study protocol for the randomized controlled SIRONA trial. Trials. 2021 Sep 28;22(1):665. doi: 10.1186/s13063-021-05631-9. PMID 34583746